CLINICAL TRIAL: NCT06871592
Title: Quantified Evaluation of Whole Face 8-points Supra-periosteum High Molecular Weight Hyaluronic Acid Injection in Asian
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Chang Cheng (Other)
Collaborators: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chang Chang Cheng, attending physician, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Other Study IDs: CMUH114-REC1-003
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Wrinkles

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Facial aging is a complex process characterized by skin atrophy, subcutaneous fat loss, and alterations in bone structure. The loss of volume, primarily due to bone resorption and loss of adjacent fat volume from different facial regions, leads to soft tissue flattening. Hyaluronic acid (HA) is a widely used biomaterial in clinical practice, known for its excellent tissue compatibility, low risk, and safety. Previous research and clinical practice have demonstrated that HA for facial lifting can help restore facial fullness, elasticity, and promote a more youthful appearance. Dermatologist previously utilized the supra-periosteum lift technique in high molecular weight hyaluronic acid injection. It was found that the material properties of high molecular weight hyaluronic acid not only made it suitable for filling but also provided lifting support, resulting in improvements in cheek fullness and facial aging. However, there has been no detailed quantitative study on the efficacy of high molecular weight hyaluronic acid for facial lifting.

To further investigate this effect, the investigators plan to conduct a prospective, open-label clinical trial. The investigators will recruit 25 adult and use an 8-point supra-periosteum facial lifting technique to inject high molecular weight hyaluronic acid. Assessments will be conducted preoperatively, postoperatively, and 4 weeks, 12 weeks and 24 weeks postoperatively to analyze the treatment efficacy. The eight injection points will be located at the brow peak, brow tail, pterion, lateral canthus, zygomatic ligament, mid-cheek, nasolabial fold, and mentalis. The investigators will use evaluation forms with four angles and six lengths, as well as the Global Aesthetic Improvement Scale, to quantify the degree of improvement in facial aging. Additionally, The investigators will use a satisfaction survey to understand subjects' perceptions of postoperative lifting effects and overall improvement satisfaction. The investigators hypothesized this study to improve facial aging in Asian patients and provide long-lasting effects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 20 and 60.
2. Subjects who are capable of understanding and comply with the study procedures, instructions, and visit schedule.
3. Subjects who voluntarily decide to participate in the entire course of the trial and provide written consent in the Informed Consent Form.

Exclusion Criteria:

1. Subjects with a history of anaphylaxis, allergy hyaluronic acid products, or any component of devices.
2. Subjects with autoimmune diseases/ received immune system and Subjects with diabetes mellitus.
3. Subjects with a history of a hypertrophic scar.
4. Pregnant or breastfeeding women.
5. Subjects with epilepsy or underlying porphyria.
6. When there is inactive disease (such as inflammation, infection or tumours) in or near the intended treatment site.
7. Treatment procedure (e.g., bioresorbable fillers, laser/light therapies, botulinum toxin A injections, face lift, facial peels, excisional facial surgery, dermal photorejuvenation clinically significant oral or maxillofacial surgery, etc.) that may interfere with the treatment area or evaluation within 6 months prior to screening as determined by the Principal Investigator.
8. The subject who received soft tissue augmentation as following at the investigational medical device injection site within 6 months prior to screening as determined by the Principal Investigator.
9. The subject who received soft tissue augmentation near the injection site with any of the following at any time.
10. Subjects with a scar or skin lesion at the investigational medical device injection site that may interfere with the judgment of the treatment effect.
11. Subjects who participated in another clinical trial within 60 days prior to screening or plan to participate in another investigation during the course of this study.
12. Subjects who plan to receive other wrinkle improvement treatment in the face during this trial.
13. Subjects who are otherwise determined by the investigator as ineligible for this study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and women aged between 20 and 60.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Eyebrow Peak angle | At Week 4, 12, and 24
  The vertices of the Eyebrow Peak angles lie at the static point eyebrow head, measured against a horizontal line parallel to the ground.
Eyebrow Tail angle | At Week 4, 12, and 24
  The vertices of the Eyebrow Tail angles lie at the static point eyebrow head, measured against a horizontal line parallel to the ground.
Pupil-Eyebrow Peak angle | At Week 4, 12, and 24
  The Pupil-Eyebrow Peak angle is then measured between this line and another line connecting nasal to eyebrow peak.
Canthus-Oral-Nasal angle | At Week 4, 12, and 24
  The Canthus-Oral-Nasal angle is measured between a line connecting oral commissure to nasal and a line connecting oral commissure to lateral canthus.
Eyebrow-Orbital length | At Week 4, 12, and 24
  The linear distances from point superior orbital rim to the inferior border of eyebrow.
Orbital-Upper Eyelid length | At Week 4, 12, and 24
  The linear distances from point superior orbital rim to the superior border of palpebral fissure.
Vertical Palpebral Fissure length | At Week 4, 12, and 24
  The size of the palpebral fissure can be determined by measuring the vertical distance between the superior and inferior borders of palpebral fissure when the eyes are at rest.
Eyebrow-Iris length | At Week 4, 12, and 24
  The horizontal distance between the lateral limbus of the iris and the eyebrow peak .
Tragus-Oral length | At Week 4, 12, and 24
  The distances between the bilateral tragi passing through the oral commissure.
Lower Facial Contouring length | At Week 4, 12, and 24
  The distances between the bilateral tragi passing through the mental protuberance.
Antiaging Scales for facial rejuvenation | At Week 4, 12, and 24
  Index 5 is identified as "neutral" or "no significant changes". Total score for the whole face was 100; either lower or higher than 50 suggesting "aging" or "rejuvenation, respectively". °: degree; mm: millimeter.

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale | At Week 4, 12, and 24
  Subjects with Global Aesthetic Improvement Scale (GAIS) from baseline after injection will be evaluated by a subjects who will judge the severity score.
  Score 0 (worse)~4 (Very much improved)